CLINICAL TRIAL: NCT05963724
Title: Efficacy of Real-Time Computer Aided-Detected of Colonic Neoplasia in an Underserved Population, A Randomized Controlled Trial
Brief Title: Real-Time CAD for Colonic Neoplasia: A RCT
Acronym: CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riverside University Health System Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 1922564-2
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
Keywords: artificial intelligence
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Real-Time Computer Aided Detection (Experimental)
  Interventions: Device: Real-Time Computer Aided Detection
- Standard Colonoscopy (Active Comparator)
  Interventions: Procedure: Stanford Colonoscopy

INTERVENTIONS:
Device: Real-Time Computer Aided Detection — This intervention involves using computer-aided detection using a real-time system (GI-Genius, Medtronic)
  Arms: Real-Time Computer Aided Detection
Procedure: Stanford Colonoscopy — This involves white-light colonoscopy
  Arms: Standard Colonoscopy

SUMMARY:
This study assesses the sensitivity and added benefits of computer-aided detection compared to standard care (white-light) in detecting colon polyps in patients undergoing colonoscopy.

DETAILED DESCRIPTION:
Failure in polyp detection leads to colon cancer after colonoscopy. Artificial intelligence systems allow real-time computer-aided detection of polyps with high-accuracy. This study will compare GI-Genius, a real-time CAD system to standard colonoscopy in terms of how many colonoscopies detect an adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing colonoscopy at RUHS
* Age > 45 years
* No contraindications to colonoscopy

Exclusion Criteria:

* Prior history of subtotal colectomy

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate | 1 year

SECONDARY OUTCOMES:
Adenomas Per Colon | 1 year
Sessile Serrated Lesion Detection Rate | 1 year
Sessile Serrated Lesions Per Colon | 1 year
False Neoplasia Rate | 1 year
Withdrawal Time | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside University Health System, Moreno Valley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thiruvengadam NR, Cote GA, Gupta S, Rodrigues M, Schneider Y, Arain MA, Solaimani P, Serrao S, Kochman ML, Saumoy M. An Evaluation of Critical Factors for the Cost-Effectiveness of Real-Time Computer-Aided Detection: Sensitivity and Threshold Analyses Using a Microsimulation Model. Gastroenterology. 2023 May;164(6):906-920. doi: 10.1053/j.gastro.2023.01.027. Epub 2023 Feb 2. PMID 36736437
- [Derived] Thiruvengadam NR, Solaimani P, Shrestha M, Buller S, Carson R, Reyes-Garcia B, Gnass RD, Wang B, Albasha N, Leonor P, Saumoy M, Coimbra R, Tabuenca A, Srikureja W, Serrao S. The Efficacy of Real-time Computer-aided Detection of Colonic Neoplasia in Community Practice: A Pragmatic Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2024 Nov;22(11):2221-2230.e15. doi: 10.1016/j.cgh.2024.02.021. Epub 2024 Mar 2. PMID 38437999